CLINICAL TRIAL: NCT06201507
Title: Efficacy and Safety of Modified BV-AVD-R Regimen in Chinese Children With Previously Untreated Intermediate- and High-risk Classical Hodgkin's Lymphoma: an Open Label, Non-randomized, Single-arm, Phase 2 Study From Single Center
Brief Title: BV-AVD-R Treatment Children Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Duan Yanlong, Assocoate chief physician, Beijing Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [2022]-E-233-Y
Record Dates: First submitted 2023-10-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Hodgkin Lymphoma
Keywords: CD30; Brentuximab vedotin; Children; Hodgkin lymphoma; Efficacy; Safety
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Rituximab; Doxorubicin; liposomal doxorubicin; Vincristine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermediate Risk (Experimental): Intermediate Risk Patients (Stage IA bulk/E, IB, IIA bulk/E, IIB, IIIA): 4 cycles of chemotherapy
  Interventions: Drug: Brentuximab vedotin; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Dacarbazine
- High Risk (Experimental): High Risk Patients (Stage IIIA bulk/ E, IIIB, IVA/B): 6 cycles of chemotherapy
  Interventions: Drug: Brentuximab vedotin; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Brentuximab vedotin — Day 1 and 15 Dose: 1.2 mg/kg/dose. (Maximum dose is 120 mg)
  Other Names: Adcetris
Drug: Rituximab — Days: 2 and 16 Dose: 375 mg/m2/dose.
  Other Names: Rituxan
Drug: Doxorubicin — Days: 1 and 15 Dose: 25 mg/m2/dose.
  Other Names: Doxil, Adriamycin
Drug: Vincristine — 1 and 15 Dose: 1.5 mg/m2/dose (max: 2 mg/dose).
  Other Names: Oncovin
Drug: Dacarbazine — 375 mg/m2 will be administered on days 1 and 15
  Other Names: DTIC

SUMMARY:
The goal of this clinical trial is to use modified Brentuximab Vedotin+doxorubicin+vinblastine+dacarbazine+Rituximab(BV-AVD-R) regimen in Chinese Classical Hodgkin's Lymphoma(HL) children. The main questions it aims to answer are:

* [Overall Response Rate(ORR) :Complete Response(CR)+Partial Response(PR)]
* [progression-free survival (PFS), event-free survival (EFS) and overall survival (OS) at 6 months and 1 year.] Participants will be given modified BV-AVD-R regimen according to rapid early responders (RER) or slow early responders (SER) after 2 cycles.

DETAILED DESCRIPTION:
This study is a prospective study with period from October 2022 to December 2024, and planned to enroll 44 children with newly diagnosed intermediate- and high-risk classical HL. All patients will undergo Positron Emission Tomography(PET)/Computed Tomography(CT) at the time of initial diagnosis and after 2 cycles of modified BV+R+AVD regimen to determine early response. Rapid early responders (RER) deﬁned as CR after 2 cycles of therapy. Slow early responders (SER) defined as no CR (partial response (PR) or stable disease) after 2 cycles of therapy. Intermediate-risk patients were stage IA bulk/E, IB, IIA bulk/E, IIB, and IIIA. High-risk patients were stage IIB bulk/E, IIIA bulk/E, IIIB, and IVA/B.

The primary endpoints include ORR (CR+PR) and adverse events. The secondary endpoints include progression-free survival (PFS), event-free survival (EFS) and overall survival (OS) at 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 18 years old, regardless of gender;
2. According to the WHO classification criteria in 2016, pathologically confirmed classic Hodgkin's lymphoma is immunohistochemical CD30 positive;
3. Newly diagnosed classic Hodgkin's lymphoma: all stages
4. The main organs function normally and meet the following definitions:

Blood routine examination: neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 75 x 109/L, hemoglobin count ≥ 80 g/dL; Liver and kidney function: AST and ALT ≤ 2.0 upper limit of normal values; Bilirubin ≤ 2.0 mg/dL; Creatinine clearance rate ≥ 60 mL/min; 5) Functional status

* For patients aged 1-16, the Lansky score is ≥ 60 points.
* For patients over 16 years old, the Karnofsky score is ≥ 60 points. 6) Previous treatment
* Except for emergency mediastinal irradiation (<1000cGy) due to superior vena cava (SVC) syndrome, Hodgkin's lymphoma guidance treatment was not allowed before.

  8) Informed consent
* Patients or their legally authorized guardians must have a thorough understanding of their illness and the nature of the study (including foreseeable risks and possible adverse reactions), and must sign an informed consent form.

Exclusion Criteria:

1. Karnofsky<60% or Lansky<60% for individuals under 16 years old.
2. Children with Hodgkin's lymphoma who have received other chemical and radiation treatments.
3. Initially rated as low-risk pediatric classic Hodgkin's lymphoma (IA, IIA, without large masses)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | Baseline up to end of randomized regimen (approximately 1 year)
  disease evaluations will be performed by PET-CT at the end of randomized regimen

SECONDARY OUTCOMES:
Progression-free survival(PFS) | 6 month and 1 year after the end of treatment
  disease evaluations will be performed at at 6 months and 1 year after the end of treatment

OTHER OUTCOMES:
Treatment Emergent Adverse Event (TEAE) | Baseline up to 30 days after last dose of study drug (approximately 1 year)
  Number of Participants Who Experience at Least One Treatment Emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Yanlong Duan, Study Chair — Beijing Children Hospital
Locations (1):
- Duan Yanlong, Beijing, China

IPD SHARING:
Plan to Share IPD: No